CLINICAL TRIAL: NCT01902316
Title: Clinical Verification for Early Diagnosis of Type 2 Diabetes Mellitus by Standard-Free, Label-Free LC-MS/MS Quantification of Glycated Peptides
Brief Title: Clinical Verification of Peptide Biomarkers for Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Beijing Institute of Technology (Other)
Responsible Party: Principal Investigator, Yulin Deng, Dean of School of Life Science, Beijing Institute of Technology
Other Study IDs: deng01
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; peptide biomarker; early diagnosis; label free
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Although diabetes has been controlled since insulin became available, it is still considered incurable and poses serious threats to human health. Reports have suggested that the hyperglycemic condition of patients with diabetes mellitus may be greatly alleviated or even reversed if it could be controlled at an early stage of diabetes. Thus, early detection and diagnosis of diabetes and prediabetes are become increasingly important in the treatment and prevention of diabetes. Diabetes mellitus is currently diagnosed by recurrent or persistent hyperglycemia. In an effort to identify novel biomarkers for diabetes, research has shown that neither plasma glucose nor glycated hemoglobin (HbA1c) levels are unable to be used in the early detection of diabetes. In this work, the investigators have found 8 biomarker candidates by developing a standard-free, label-free MS-based proteomics method based on standard protein (human serum albumin, the highest abundance protein in human plasma) model in vitro. Then, the investigators wanted to verify these biomarker candidates by clinical plasma samples to see if there is significant quantitative difference between normal people and diabetes patients.

DETAILED DESCRIPTION:
The procedure of clinical study was:

1. to get plasma samples from hospital;
2. digestion of plasma protein-mixture by trypsin;
3. run mass spectrometry and monitor the amount of target HSA-peptides.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus cases;
* Impaired Glucose Tolerance cases;
* Normal Glucose Tolerance cases

Exclusion Criteria:

* Type 1 Diabetes Mellitus cases;
* Gestational Diabetes Mellitus cases;
* Hepatitis patients

Ages: 35 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: university hospital, plasma samples of physical examination, faculties and staff of a certain university
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
measurement of the amount of plasma peptides | two years
  The investigators have found 8 biomarker candidates by developing a standard-free, label-free MS-based proteomics method based on standard protein (human serum albumin, the highest abundance protein in human plasma) model in vitro. Then, the investigators wanted to verify these biomarker candidates by clinical plasma samples to see if there is significant quantitative difference between normal people and diabetes patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yulin Deng, Ph.D., Principal Investigator — School of Life Science, BIT